CLINICAL TRIAL: NCT03466619
Title: Assessment of Safety and Efficacy of Inflatable Penile Prothesis in Patients With Erectile Dysfunction
Brief Title: Penile Prosthesis in Patients With Erectile Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Khaled Hafez
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Penile Prosthesis

STUDY DESIGN:
Intervention Model Description: inflatable penile prosthesis (IPP)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inflatable penile prosthesis (IPP) (Experimental): inflatable penile prosthesis (IPP)
  Interventions: Device: inflatable penile prosthesis (IPP)

INTERVENTIONS:
Device: inflatable penile prosthesis (IPP) — inflatable penile prosthesis (IPP)
  Other Names: penile prosthesis (IPP)

SUMMARY:
Erectile dysfunction (ED) is defined as the persistent inability to attain and or maintain an erection sufficient to permit satisfactory sexual performance

DETAILED DESCRIPTION:
In the literature, well- designed studies evaluating safety and efficacy of inflatable penile prosthesis (IPP) is lacking. So, this series aimed at investigating this prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of ED with contraindication or failure of medical treatment

Exclusion Criteria:

* Patients lacking manual dexterity or mental abilities necessary to operate the pump
* General contraindications as uncorrectable bleeding tendency

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 100 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved erectile dysfunction | 3 years
  The number of patients with improved erectile dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mohamed Hafez Morsy Almekaty, Msc, Principal Investigator — Urology Department- Tanta University; Samir Abdelhakim Elgamal, Prof, Principal Investigator — Urology Department- Tanta University; Suks Minhas, Prof, Principal Investigator — Professor of urology University College London Hospital(UCLH)London, UK
Locations (1):
- Tanta university - faculty of medicine, Cairo, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided